CLINICAL TRIAL: NCT06125899
Title: Intervention for Depression in Underserved Geriatric Populations
Brief Title: Protocol for a Feasibility Cluster Randomised Controlled Trial of a Home-based Depression Care for Older People Delivered by Lay Providers in Nigeria
Acronym: INDIGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, Akin Ojagbemi, Senior Lecturer, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 220684/Z/20/Z
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Depression in Old Age

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Age emhGAP-IG (Experimental): * Adapted emhGAP-IG;
  * Adapted Problem-Solving Therapy (PST-PC)
  * Support/supervision of lay providers
  * Links to social support resources.
  Interventions: Behavioral: emhGAP-Age
- Generic emhGAP-IG (Active Comparator): Psychoeducation and stress reduction
  Interventions: Behavioral: emhGAP-Age

INTERVENTIONS:
Behavioral: emhGAP-Age — * Adapted emhGAP-IG;
  * Adapted Problem-Solving Therapy (PST-PC)
  * Support/supervision of lay providers
  * Links to social support resources.

SUMMARY:
The aim of this hybrid (Effectiveness-Implementation) cluster randomised controlled clinical trial is to test the feasibility of implementing an age-appropriate electronic version of the WHO Mental Health Gap Action Programme Intervention Guide (emhGAP-Age) in routine home-based care of older Nigerians with depression. The main questions it aims to answer are:

1. Whether the emhGAP-Age demonstrate sufficient signals of effectiveness in the identification and home management of late life depression to permit for further exploration in a fully powered clinical trial?
2. What are the logistical, programmatic, and operational requirements for a home-delivered emhGAP-Age in a sample of older people with depression in Nigeria? Consenting older participants with depression in the intervention arm will receive treatment based on emhGAP-Age which consists of;

   * Adapted electronic generic version of the WHO Mental Health Gap Action Programme Intervention Guide (emhGAP-IG)
   * Adapted Problem-Solving Therapy (PST-PC)
   * Support/supervision of providers
   * Links to social support resources. Researchers will compare with treatment based on the basic specification in the generic emhGAP-IG (consisting of basic psychoeducation and stress reduction) for effects on depression remission.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years,
2. PHQ-9 score of ≥11 during routine consultation

Exclusion Criteria:

1. Severe co-morbidity requiring urgent attention.
2. Severe cognitive impairment/dementia (Community Screening Instruments for Dementia score≤ 20) .
3. Active suicidal intention.
4. Evidence of bipolar/psychosis/severe substance use disorders.
5. Planning to move out of the study catchment area within 6 months.
6. Refusing/lacking capacity to consent/accent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Depression remission | At six months post trial entry
  Patient Health Questionnaire (PHQ-9) score < 6